CLINICAL TRIAL: NCT03673956
Title: Topical Antibiotics in Chronic Rhinosinusitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Garret W. Choby, Senior Associate Consultant - Department of Otorhinolaryngology; Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-006599
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Mupirocin; Tobramycin; Levofloxacin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mupirocin Topical Antibiotic Nasal Saline Rinse (Experimental): Subjects with a history of chronic rhinosinusitis (CRS) who had previously undergone endonasal sinus surgery (minimum of maxillary antrostomy and anterior ethmoidectomy), will receive a trial of Mupirocin topical antibiotic rinses. Subjects will undergo a baseline assessment including an aerobic sinus bacterial culture with antibiotic sensitivity to determine baseline microbial antibiotic resistance and to direct selection of appropriate topical antibiotic therapy.
  Interventions: Drug: Mupirocin
- Tobramycin Topical Antibiotic Nasal Saline Rinse (Experimental): Subjects with a history of chronic rhinosinusitis (CRS) who had previously undergone endonasal sinus surgery (minimum of maxillary antrostomy and anterior ethmoidectomy), will receive a trial of Tobramycin topical antibiotic rinses. Subjects will undergo a baseline assessment including an aerobic sinus bacterial culture with antibiotic sensitivity to determine baseline microbial antibiotic resistance and to direct selection of appropriate topical antibiotic therapy.
  Interventions: Drug: Tobramycin
- Levofloxacin Topical Antibiotic Nasal Saline Rinse (Experimental): Subjects with a history of chronic rhinosinusitis (CRS) who had previously undergone endonasal sinus surgery (minimum of maxillary antrostomy and anterior ethmoidectomy), will receive a trial of Levofloxacin topical antibiotic rinses. Subjects will undergo a baseline assessment including an aerobic sinus bacterial culture with antibiotic sensitivity to determine baseline microbial antibiotic resistance and to direct selection of appropriate topical antibiotic therapy.
  Interventions: Drug: Levofloxacin
- Vancomycin Topical Antibiotic Nasal Saline Rinse (Experimental): Subjects with a history of chronic rhinosinusitis (CRS) who had previously undergone endonasal sinus surgery (minimum of maxillary antrostomy and anterior ethmoidectomy), will receive a trial of Vancomycin topical antibiotic rinses. Subjects will undergo a baseline assessment including an aerobic sinus bacterial culture with antibiotic sensitivity to determine baseline microbial antibiotic resistance and to direct selection of appropriate topical antibiotic therapy.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Mupirocin — 30mg capsules dissolved in a standard 240mL saline irrigation rinse and self-administered through nasal saline irrigation twice per day over 30 days.
  Arms: Mupirocin Topical Antibiotic Nasal Saline Rinse
Drug: Tobramycin — 240mg capsules dissolved in a standard 240mL saline irrigation rinse and self-administered through nasal saline irrigation twice per day over 30 days.
  Arms: Tobramycin Topical Antibiotic Nasal Saline Rinse
Drug: Levofloxacin — 240mg capsules dissolved in a standard 240mL saline irrigation rinse and self-administered through nasal saline irrigation twice per day over 30 days.
  Arms: Levofloxacin Topical Antibiotic Nasal Saline Rinse
Drug: Vancomycin — 240mg capsules dissolved in a standard 240mL saline irrigation rinse and self-administered through nasal saline irrigation twice per day over 30 days.
  Arms: Vancomycin Topical Antibiotic Nasal Saline Rinse

SUMMARY:
Researchers are trying to find out if patients develop antibiotic resistant organisms after the use of topical antibiotics in the treatment of chronic rhinosinusitis.

DETAILED DESCRIPTION:
There is a certain group of patients that has chronic rhinosinusitis that has continued even with treatment including saline and steroid nasal irrigations as well as oral steroids and antibiotics and surgery.

In these patients, the use of topical antibiotic nasal rinses may be of benefit to their disease. The use of topical antibiotic nasal rinses is commonly used as standard of care already throughout the country for refractory chronic rhinosinusitis including here at the Mayo Clinic. Our pharmacy has compounded this medication for this specific purpose. As such, this study is not aimed at a 'novel medication', but rather to investigate the efficacy of a medication already in common use but without great evidence.

The investigators are doing this research study to find out if patients develop antibiotic resistant organisms after the use of topical antibiotics in the treatment of chronic rhinosinusitis.

In addition, this study will look at the effects of topical antibiotics on patient symptoms as measured by a patient survey called the Sino-Nasal Outcomes Test (SNOT-22) and in-office an exam of the inside of their nose, including with a scope (a camera on the end of a long tube).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18-80 years old, diagnosed with chronic rhinosinusitis who have undergone previous functional endoscopic sinus surgery including at minimum maxillary antrostomy and anterior ethmoidectomy
* Active mucopurulence on endoscopic examination with corresponding culture demonstrating pathogenic bacterial growth
* Completion of written informed consent
* No prior enrollment into this study
* Refractory to maximal medical therapy

Exclusion Criteria:

* Patient has not had prior endoscopic sinus surgery consisting of at minimum maxillary antrostomy and anterior ethmoidectomy
* Patient is currently being treated with oral antibiotics
* Patient has been treated with oral or topical antibiotics within the past 14 days
* Participation in an investigational drug study simultaneously with participation in this study
* Concurrent use of oral steroids
* Allergy to Tobramycin, Mupirocin, Gentamicin and Levofloxacin
* Known to currently be pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garret W Choby, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Mupirocin Antibiotic Nasal Saline Rinse: Subjects with a history of chronic rhinosinusitis (CRS) who had previously undergone endonasal sinus surgery (minimum of maxillary antrostomy and anterior ethmoidectomy), will receive a trial of Mupirocin topical antibiotic rinses. Subjects will undergo a baseline assessment including an aerobic sinus bacterial culture with antibiotic sensitivity to determine baseline microbial antibiotic resistance and to direct selection of appropriate topical antibiotic therapy.
  Mupirocin: 30mg capsules dissolved in a standard 240mL saline irrigation rinse and self-administered through nasal saline irrigation twice per day over 30 days.
Period: Overall Study
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse
Started | 12 | 1 | 5 | 1
Completed | 10 | 1 | 5 | 1
Not Completed | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Did not use the prescribed topical antibiotics as directed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse | Total
Number analyzed (Participants) | 12 | 1 | 5 | 1 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 7 | 0 | 2 | 0 | 9
  >=65 years | 4 | 1 | 3 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 4 | 1 | 12
  Male | 5 | 1 | 1 | 0 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 1 | 5 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Subjects Who Developed Antibiotic Resistance Organisms
Description: Number of subjects who developed new antibiotic resistance organisms measured by nasal swab of the affected sinonasal cavity and sent for stain, culture, and sensitivity.
Time Frame: Post-intervention (within 21 days of intervention completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse
Number analyzed (Participants) | 10 | 1 | 5 | 1
Participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Change in Patient Symptoms as Measured by the Sino-Nasal Outcomes Test (SNOT-22) Survey
Description: Scores are measured from 0-5 in a 22-item validated survey. Total scores range from 0-110 with higher scores indicating greater burden of sinonasal symptoms.
Time Frame: Baseline, Post-intervention (within 21 days of intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse
Number analyzed (Participants) | 8 | 1 | 2 | 1
units on a scale | -18 (21.8) | 14 | -25.5 (34.6) | -11

3. Secondary Outcome: Change in Patient Physical Exam as Measured by the Lund-Kennedy Endoscopic Exam Scores.
Description: Scores are measured on a 0-2 scale for nasal polyps, edema, and secretions in both right and left nasal cavities. Total scores range from 0 to 12 with higher scores indicating greater evidence of sinonasal disease on physical exam.
Time Frame: Baseline, Post-intervention (within 21 days of intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse
Number analyzed (Participants) | 10 | 1 | 5 | 1
units on a scale | -5.3 (2.8) | -3 | -2.4 (2.4) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 2 months on all participants.
Arm/Group | Mupirocin Antibiotic Nasal Saline Rinse | Tobramycin Topical Antibiotic Nasal Saline Rinse | Levofloxacin Topical Antibiotic Nasal Saline Rinse | Vancomycin Topical Antibiotic Nasal Saline Rinse
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/1 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 0/12 | 1/1 | 1/5 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mupirocin Antibiotic Nasal Saline Rinse (N=12) | Tobramycin Topical Antibiotic Nasal Saline Rinse (N=1) | Levofloxacin Topical Antibiotic Nasal Saline Rinse (N=5) | Vancomycin Topical Antibiotic Nasal Saline Rinse (N=1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Face Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial Pressure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Drainage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03673956/Prot_SAP_000.pdf